CLINICAL TRIAL: NCT00502814
Title: 3-Dimensional Form and Soft Tissue Biomechanics of the Breast
Status: Terminated | Type: Observational
Why Stopped: Sample size too small for data analysis.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID01-305
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; 3-D Optical Surface Scan; Soft Tissue Biomechanics; Mechanical Testing; Skin Ultrasound; Magnetic Resonance Imaging; CT Scan
MeSH Terms: conditions — Breast Neoplasms | interventions — Mechanical Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Breast Cancer.
  Interventions: Procedure: 3-D Optical Surface Scan; Procedure: Mechanical Testing; Procedure: Cutaneous Ultrasound; Procedure: Breast MRI and/or CT

INTERVENTIONS:
Procedure: 3-D Optical Surface Scan — 3-D digitized images of the breasts and chest will be taken over a period of five minutes.
Procedure: Mechanical Testing — A small device with a mild suction will be used to measure how the skin tends to stretch.
Procedure: Cutaneous Ultrasound — Cutaneous ultrasound using a 20 MHz machine and the skin thickness will be recorded.
Procedure: Breast MRI and/or CT — Imaging of the breasts and chest using an MRI and/or CT scan over about one hour.

SUMMARY:
The goal of this clinical research study is to characterize the 3-dimensional form and mechanical properties of the breast. Researchers want to do this in order to develop new high technology tools for improving the diagnosis and treatment of breast cancer in women.

DETAILED DESCRIPTION:
Patients who participate in the study will have general physical and demographic information recorded. Height, weight, age, race, menstrual status, and bra size will all be recorded. Patients will have a breast physical exam. Researchers will then perform several painless tests and imaging studies to evaluate the mechanical properties of the skin and the shape and tissue composition of the breasts.

Patients in this study will go through a series of evaluations as listed below.

1. 3-D Optical Surface Scan (estimated time required: 5 minutes) The camera system with a safe scanning laser will be used to take 3-D digitized images of the breasts and chest. Multiple images may be necessary to get a complete rendering of both breasts. Each image requires less than 0.6 seconds to take. This process is similar to the routine photography currently performed on most patients.
2. Mechanical testing (estimated time required: 1 hour) A small device will be applied with the surface of the skin at several locations on the breasts. A mild suction will be applied for several seconds for each measurement. This will measure how the skin tends to stretch. The instruments used are very sensitive and provide the information needed with very small, painless amounts of movement in the skin. In addition to evaluating characteristics of the breast skin, one additional measure will be taken on the skin at the front of the forearm area to help understand your general skin qualities.
3. Skin Ultrasound (estimated time required: 15 minutes) Patients will have a cutaneous ultrasound using the 20 MHz machine and the skin thickness will be recorded in each of the domains. A trained technician will complete this exam. In addition to evaluating characteristics of the breast skin, one additional measure will be taken on the skin at the front of the forearm area to help understand your general skin qualities.
4. Breast MRI and/or CT (estimated time required: 1 hour) Some patients will be scheduled for imaging of the breasts and chest using MRI and/or CT. These images will be taken free-of-charge as they are not required for standard of care.

Participation will be over once the evaluations are complete.

This is an investigational study. A total of 200 patients will take part in this study. All will be enrolled at M. D. Anderson. After the first 50 patients are enrolled, the results will be studied to see if the study will continue. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Greater than 18 years old.
3. Presenting complaint requires breast physical examination.
4. Free of connective tissue disorders and cutaneous malignancy on the breast.
5. Free of medical conditions that contraindicate MRI or CT scanning.
6. Willing to participate in the study and able to complete informed consent.

Exclusion Criteria:

1) Patients who do not meet inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Breast Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2003-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Individual 3-dimensional Form and Mechanical Properties of Patient's Breast | Patient participation is approximately 1 Day for breast scans and mechanical measure, as well as ultrasound and Breast MRI/CT

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Beahm, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org